CLINICAL TRIAL: NCT06780124
Title: An Exploratory Randomized, Double-Blind, Placebo-Controlled, First-in-Human Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of ZE63-0302 in Healthy Volunteers
Brief Title: Сlinical Study Aiming to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of ZE63-0302 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eilean Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ZE63-0302-0001
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Acute leukemia; Acute KMTRAR mutated myeloid leukemia; Acute NPM1 mutated myeloid leukemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Level 1 Single dose (Experimental): Dose level 1: 6 participants will receive 20 mg ZE63-0302 and 2 participants will receive placebo under fasted conditions.
  Interventions: Drug: ZE63-0302 or placebo
- Level 2 Single dose (Experimental): Dose level 2: 6 participants will receive 100 mg ZE63-0302 and 2 participants will receive placebo under fasted conditions.
  Interventions: Drug: ZE63-0302 or placebo
- Level 3 Single dose (Experimental): Dose level 3: 6 participants will receive 300 mg ZE63-0302 and 2 participants will receive placebo under fasted conditions.
  Interventions: Drug: ZE63-0302 or placebo
- Level 4 Single dose (Experimental): Dose level 4: 6 participants will receive 600 mg ZE63-0302 and 2 participants will receive placebo under fasted conditions.
  Interventions: Drug: ZE63-0302 or placebo
- Level 5 Single dose (Experimental): Dose level 5: 9 participants will receive 300 mg ZE63-0302 and 3 participants will receive placebo under fed conditions.
  Interventions: Drug: ZE63-0302 or placebo
- Level 6 Single dose (Experimental): Dose level 6: 6 participants will receive 600 mg ZE63-0302 plus itraconazole and 2 participants will receive placebo plus itraconazole under fasted conditions.
  Interventions: Drug: ZE63-0302 or placebo
- Level 7 Single dose (Experimental): Dose level 7: 3 participants will receive 600 mg ZE63-0302 and 1 participant will receive placebo under fed conditions.
  Interventions: Drug: ZE63-0302 or placebo
- Level 1 Multiple doses (Experimental): Dose level 1: 6 participants will receive 600 mg ZE63-0302 and 2 participants will receive placebo once daily under fasted and/or fed conditions. Duration of dosing (ZE63-0302 or placebo) is 7 days.
  Interventions: Drug: ZE63-0302 or placebo
- Level 2 Multiple doses (Experimental): Dose level 2: 6 participants will receive 300 mg ZE63-0302 and 2 participants will receive placebo twice daily under fasted and/or fed conditions. Duration of dosing (ZE63-0302 or placebo) is 7 days.
  Interventions: Drug: ZE63-0302 or placebo

INTERVENTIONS:
Drug: ZE63-0302 or placebo — The participants will receive ZE63-0302 or placebo

SUMMARY:
A first-in-human study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple ascending doses of ZE63-0302 administered orally in healthy volunteers.

DETAILED DESCRIPTION:
This is an exploratory Phase I, single- and multiple-dose escalation clinical trial conducted in healthy volunteers. The safety, tolerability, pharmacokinetics and pharmacodynamics of ZE63-0302 following oral administration in healthy volunteers will be evaluated using a randomized, double-blind, placebo-controlled trial design.

This study will be subdivided into two parts: a single ascending dose (SAD) part and a multiple ascending dose (MAD) part.

Healthy volunteers (BMI ≥ 18.5 and ≤ 32.0 kg/m2) and healthy volunteers with a high BMI (≥ 30.0 and ≤ 35.0 kg/m2) will be enrolled to receive single ascending doses (SAD) of ZE63-0302 or placebo under fasted or fed conditions, depending on the cohort, and healthy volunteers (BMI ≥ 18.5 and ≤ 32.0 kg/m2) will receive multiple ascending doses (MAD) of ZE63-0302 or placebo under fasted or fed conditions, depending on the cohort. The starting dose will be 20 mg with up to 7 SAD and 4 MAD cohorts planned. Sentinel dosing will be utilized in SAD Cohorts 1 to 4.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 55 years of age (inclusive) at screening.
3. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2, with a body weight (to 1 decimal place) ≥ 50.0 kg at screening, to be included in the main group for all SAD and MAD cohorts. BMI ≥ 30.0 and ≤ 35.0 kg/m2, with a body weight (to 1 decimal place) ≥ 50.0 kg at screening, to be included in the high BMI group for SAD Cohorts 5 and 7.
4. Medically healthy without clinically significant abnormalities (in the opinion of the Investigator) at the screening visit and prior to dosing at the timepoints indicated in the SoA, including:

   1. Physical examination without any clinically significant findings.
   2. Systolic blood pressure in the range of 90 mm Hg to 140 mm Hg; diastolic blood pressure in the range of 40 mm Hg to 90 mm Hg.
   3. HR in the range of 40 to 100 bpm after at least 5 minutes in a supine position
   4. Body temperature (tympanic or oral) in the range 35.5°C to 37.5°C (inclusive).
   5. No clinically significant findings in serum chemistry, hematology, coagulation and urinalysis tests as judged by the Investigator. Note: for SAD Cohort 6, ALT, AST, ALP and gamma-glutamyl transferase (GGT) must be normal (within the reference range).
   6. Triplicate 12-lead ECG (taken after the volunteer has been supine for at least 5 minutes) with a QTcF ≤ 450 msec for males and ≤ 470 msec for females and no clinically significant abnormalities.
5. Be nonsmokers (including tobacco, nicotine replacement therapy, e-cigarettes and marijuana) for at least 3 months prior to first study drug administration (self-reported to the Investigator) at screening visit, Day -4 (SAD Cohort 6 only) and at check-in on Day -1.
6. Female volunteers must:

   1. Be of nonchildbearing potential i.e., surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before screening) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause, and a follicle-stimulating hormone (FSH) level >40 IU/L at the screening visit), or
   2. If of childbearing potential, must agree not to donate ova, not to attempt to become pregnant and, if engaging in sexual intercourse with a male partner, must agree to use an acceptable method of contraception from one month prior to screening until at least 30 days after the last dose of study drug.
7. Male volunteers must agree not to donate sperm and, if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use an acceptable method of contraception from signing the consent form until at least 90 days after the last dose of study drug.
8. Have suitable venous access for blood sampling.
9. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or major surgery within the past 3 months determined by the PI to be clinically significant.
2. Acute infections or infestations within 4 weeks prior to dosing or current infection that requires systemically absorbed antibiotic, antifungal, antiparasitic or antiviral medications.
3. Presence or history of any abnormality or illness, including gastrointestinal surgery, which in the opinion of the PI may affect absorption, distribution, metabolism or elimination of the study drug.
4. Any history of malignant disease in the last 5 years (excludes surgically resected skin squamous cell or basal cell carcinoma).
5. Any screening laboratory result outside the normal laboratory reference range (as confirmed upon repeated testing) and deemed clinically significant by the PI.

   Participants who have Gilbert's syndrome, or who have hyperbilirubinemia consistent with Gilbert's syndrome, will not be eligible.
6. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia.
7. Use of or plans to use systemic immunosuppressive (e.g., corticosteroids by any route, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (e.g., interferon) within 5 half-lives of individual agent or within 28 days (whichever is longer) prior to dosing or during the study.
8. Use of or plans to use agents (e.g., grapefruit and grapefruit products) that have clinically significant interaction with CYP3A4 or the use of any medications that could have a significantly impact on organ function (e.g., barbiturates, omeprazole, cimetidine) during the study or within 5 half-lives of individual agent or within 28 days (whichever is longer) prior to dosing.
9. History of risk factors for torsade de pointes (including a family history of long QT syndrome or sudden cardiac death) or clinically significant arrythmia.
10. Participant is planning to have surgery between Screening and the EoS visit.
11. Positive test results for active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies at the screening visit.
12. Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
13. Estimated creatinine clearance < 60 mL/min using the Cockcroft-Gault formula.
14. History of any drug or alcohol abuse in the past 2 years defined as >21 units of alcohol per week for males and >14 units of alcohol per week for females. Where 1 unit = 360 mL of beer, 150 mL wine, or 30 mL of spirits.
15. No alcohol consumption within 24 hours prior to Day -4 (SAD Cohort 6 only), and/or check-in (Day -1).
16. Positive drugs of abuse, cotinine or alcohol breath test results at the screening visit, Day -4 (SAD Cohort 6 only) or at check-in (Day -1).
17. Use of any prescription medications within 14 days or at least 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, including oral contraceptives and use of any over-the-counter medication (including herbal products, nutritional, diet aids, vitamin supplements, minerals and hormone supplements) within 7 days or at least 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, with the exception of the occasional use of paracetamol (doses of 500 mg up to every 6 hours or 2 g per day maximum for no more than 3 consecutive days).
18. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the Investigator, would interfere with thevolunteer's ability to participate in the trial
19. Known hypersensitivity to any of the study drug ingredients.
20. Use of any inactivated vaccinations within 14 days, or any live vaccinations within 30 days prior to the first study drug administration. Note: Subjects vaccinated for COVID-19 or influenza within at least 2 weeks prior to enrollment or earlier will be considered eligible for enrollment as long as they do not present with post-vaccination clinical symptoms, have a negative rapid antigen test (in the case of COVID-19), and are deemed otherwise healthy.
21. For women of childbearing potential, a positive serum pregnancy test at the screening visit or a positive urine pregnancy test (with confirmatory serum pregnancy test) at check-in (Day -1).
22. Females who are breastfeeding or planning to breast feed at any time during the study.
23. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to first study drug administration, or receipt of a blood transfusion within 1 year of first study drug administration.
24. Receiving an investigational drug in another clinical trial within 60 days or 5 half-lives of the investigational agent (whichever is longer) prior to the first study drug administration.
25. Any other condition or prior therapy that in the opinion of the Investigators would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.
26. Any history of long COVID infection (defined by continuation or development of new symptoms 3 months after the initial SARS-CoV-2 infection, with these symptoms lasting for at least 2 months with no other explanation).

    Additional exclusion criteria for SAD Cohort 6 only:
27. History or presence of clinically significant hypersensitivity or idiosyncratic reaction to itraconazole or other azole compounds, or any inactive ingredients.
28. History or presence of clinically significant liver disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics of ZE63-0302 | Within 15 min prior to dosing with ZE63-0302/placebo to 168 hours post-dose for SAD . Within 15 min prior to dosing with ZE63-0302/placebo to 264 hours post-dose for MAD.
  Plasma concentration, ng/mL
Effect of BMI on the PK of ZE63-0302 in plasma following administration of single oral doses (for dose levels 5 and 6 only) | Within 15 min prior to dosing with ZE63-0302/placebo to 168 h post-dose.
  Plasma concentration, ng/mL

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | From the signing of the consent form until day 8 for SAD dose levels 1-5 and 7 and until day 11 for SAD dose level 6 and until day 18 for MAD.
  Incidence of AEs/SAEs (serious adverse events)including significant changes from baseline in body weight, vital signs, electrocardiogram parameters and laboratory assessments qualifying and reported as AEs.

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research Ltd, Perth, Nedlands, Australia

IPD SHARING:
Plan to Share IPD: Undecided